CLINICAL TRIAL: NCT06292039
Title: Identifying & Addressing Unmet Needs of Injury Survivors at a Safety Net Hospital in San Francisco
Brief Title: Human-centered Injury Thrivorship Pathway for Survivors of Physical Trauma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: P0555788; 2KL2TR001870 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-03-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Injury Traumatic; Survivorship; Trauma Injury
Keywords: Social determinants of health; Community-engaged research; Unmet needs
MeSH Terms: conditions — Wounds and Injuries; Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injury Thrivorship Pathway (Experimental): Enrollment in the human-centered injury thrivorship pathway.
  Interventions: Other: Human-Centered Injury Thrivorship Pathway

INTERVENTIONS:
Other: Human-Centered Injury Thrivorship Pathway — Enrollment in the human-centered injury thrivorship pathway.

SUMMARY:
The goal of this clinical trial is to pilot and evaluate a human-centered injury thrivorship pathway in injury survivors. The main question it aims to answer is:

• Is the pathway appropriate, acceptable, and feasible to meet the medical and social needs of injury survivors?

Injury survivors will be purposively sampled to enroll in the pathway and asked to participate in in-depth interviews and their use of pathway resources will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old presenting with a physical injury to Zuckerberg San Francisco General Hospital
* Admitted to the hospital ≥ 24 hours
* Discharged from the hospital alive
* San Francisco resident or unhoused in San Francisco
* Capacity for informed consent

Exclusion Criteria:

* Patient < 18 years old
* Deceased during index hospitalization
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Early Implementation Outcomes - Acceptability, Appropriateness, Feasibility | 8-12 weeks post-pathway enrollment
  Early implementation outcomes will be assessed via purposive sampling of pathway participants, their caregivers, and trauma care stakeholders for in-depth semi-structured interviews. "Acceptability is the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Appropriateness is the perceived fit, relevance, or compatibility of the innovation or evidence based practice for a given practice setting, provider, or consumer; and/or perceived fit of the innovation to address a particular issue or problem. Feasibility is defined as the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting."

SECONDARY OUTCOMES:
Participant pathway resource utilization - type | 8-12 weeks post-pathway enrollment plus subsequent time points if continued resource engagement until study completion up to 1 year
  Participant engagement with applicable pathway resources will be tracked by type of resource(s) accessed
Participant pathway resource utilization - frequency | 8-12 weeks post-pathway enrollment plus subsequent time points if continued resource engagement until study completion up to 1 year
  Participant engagement with applicable pathway resources will be tracked by frequency of use of the resource(s)
Participant pathway resource utilization - duration | 8-12 weeks post-pathway enrollment plus subsequent time points if continued resource engagement until study completion up to 1 year
  Participant engagement with applicable pathway resources will be tracked by duration of use of the resource(s)
Participant pathway resource utilization - % utilized | 8-12 weeks post-pathway enrollment plus subsequent time points if continued resource engagement until study completion up to 1 year
  Participant engagement with applicable pathway resources will be tracked by overall % of resources utilized out of resource(s) offered

CONTACTS AND LOCATIONS:
Overall Officials: Marissa A Boeck, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
The investigators are undecided how individual participant data will be shared with other researchers, which the investigators will update prior to the initial recruitment date. The primary outcome will be qualitative data from in-depth semi-structured interviews linked to participant demographic and clinical information. The secondary outcome will be quantitative based on resource utilization, also linked to participant demographic and clinical information.

REFERENCES:
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426